CLINICAL TRIAL: NCT05614115
Title: Safety, Tolerability, and Feasibility of Empagliflozin Therapy in Dialysis-dependent ESKD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Monique Cho, Associate Professor in the Department of Medicine, Division of Nephrology & Hypertension, University of Utah
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00155825; 1R01DK131265 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2022-11-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: End-stage Kidney Disease; Kidney Disease, Chronic; Dialysis; Diabetic; Non-diabetic; Kidney Dysfunction; Kidney Failure; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two phases, a dose-escalation phase (week 0-4) and a treatment phase (week 5-12).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Empagliflozin 10mg (Experimental): Empagliflozin10mg oral: Those randomized to 10 mg daily dose will be treated with 10 mg QD throughout the dose escalation and the treatment phase for a total of 12 weeks.
  Interventions: Drug: Empagliflozin
- Empagliflozin 25mg (Experimental): Empagliflozin 25 mg oral: Those randomized to 25 mg daily dose will be treated with 10 mg QD for the first 2 weeks before escalating the dose to 25 mg QD in week 3, based on tolerability. At the end of the dose-escalation phase (weeks 3-4), participants will continue the randomized assignment for additional 8 weeks (weeks 5-12, treatment phase), for a total of 12 weeks.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Encapsulated placebo with an identical appearance to empagliflozin: Those randomized to placebo will be treated with an oral placebo QD throughout the dose escalation and the treatment phase for a total of 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin — is a sodium-glucose co-transporter 2 (SGLT2) inhibitor.
  Other Names: Jardiance®; CL-JAR-100113 02.28.2022
  Arms: Empagliflozin 10mg; Empagliflozin 25mg
Other: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if empagliflozin, a new diabetic medication that has been shown to be very effective in lowering the risk of heart failure, is safe and tolerated in dialysis patients. In the recent years, empagliflozin has become a major tool to prevent heart failure hospitalization and to reduce the risk for cardiovascular death in diabetic and non-diabetic patients. Although patients with severe chronic kidney disease and ESKD have very high risk of heart failure and cardiovascular death, they have been excluded from all of the previous studies. If this medication is found to be well tolerated and safe in dialysis patients through this study, future clinical studies can evaluate if this medication can also reduce the risk of heart failure and cardiovascular death in dialysis patients.

DETAILED DESCRIPTION:
Patients on dialysis have a very high risk of heart failure and heart-related death compared to people who do not require dialysis. While treatment options for heart failure have improved over the years for those without kidney disease, there has been very limited discoveries to improve survival for dialysis patients.

Empagliflozin, a new diabetic medication that works by making the kidney put out more sugar in the urine, has recently shown to have significant efficacy to protect the kidney and to reduce heart failure hospitalization and cardiovascular death in both diabetic and non-diabetic patients. Studies suggest that this medication may have benefits on the heart, fat cells, blood vessels, and possibly other organ systems. The benefit remains consistent whether you have diabetes or not. Empagliflozin is now approved by the U.S. Food and Drug Administration (FDA) to treat not only diabetes but also chronic kidney disease and to reduce the risk of cardiovascular death and hospitalization for heart failure in adults regardless of the diabetes status.

The clinical studies, however, have excluded those with severe kidney disease and those requiring dialysis. The safety of empagliflozin in the dialysis patients has not been established, and thus it is not available for people with end-stage kidney disease. If empagliflozin is safe in dialysis patients, it may potentially become a very powerful tool to lower the risk of heart-related complications and prolong survival.

Although empagliflozin is approved by the FDA to treat patients with chronic kidney disease, heart failure, and/or diabetes, our study will evaluate empagliflozin as an investigational drug to assess if it is safe in patients receiving chronic dialysis. If we can establish safety, the next step would be to conduct a larger clinical study to evaluate its ability to lower heart failure and death risk in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* include diabetic and non-diabetic adults
* dialysis treatment history of ≥3 months

Exclusion Criteria:

* type 1 diabetes
* ongoing intravenous antibiotic therapy for infectious disease
* active treatment for malignancy
* unhealed lower extremity skin ulceration
* history of Fournier's gangrene
* diabetic ketoacidosis
* severe hypoglycemia (requiring external assistance within the past one year)
* allergy to empagliflozin
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
The proportion of participants in each intervention group who remain in follow-up and adhere to the full randomized dose of empagliflozin at the end of the 12-week intervention period. | 12 weeks

SECONDARY OUTCOMES:
Proportions of participants in each group who reduce and/or discontinue treatment for safety | 12-weeks
  Safety outcomes (to be assessed in each treatment group):
  1. Proportions of participants with any of the following prespecified adverse events of interest: (i) Severe hypoglycemia1; (ii) Ketoacidosis; (iii) Hypotension; (iv) Genital infection; (v) Hepatic injury
  2. Composite of the individual components of the prespecified adverse events of interest (i) through (v)
  3. Occurrence of any hospitalization and/or visit to Emergency Department
Proportions of participants in each group who reduce and/or discontinue treatment because of intolerance (i.e., allergy, nausea) or other reasons unrelated to safety (i.e., pill burden, study withdrawal due to transplant) | 12-weeks
Proportions of participants in each group who have ≥ 80% pill count compliance. | 12-weeks
Dialytic clearance of empagliflozin | 4 hours post-dose during hemodialysis
Long-term accumulation of empagliflozin | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No